CLINICAL TRIAL: NCT04518228
Title: Pharmacokinetic Properties of Antiretroviral and Anti-Tuberculosis Drugs During Pregnancy and Postpartum
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry); ViiV Healthcare (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2026; 38609 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-03-05; First posted 2020-08-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — bictegravir; tenofovir alafenamide; cabotegravir; dolutegravir; atazanavir, ritonavir drug combination; Darunavir; Ritonavir; Lopinavir; Cobicistat; doravirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Component 1: Arm 1.1: Bictegravir (BIC) 50 mg q.d.: Women ≥ 20 weeks gestation not receiving TB drugs and receiving bictegravir (BIC) 50 mg once daily (q.d.), and their infants
  Interventions: Drug: Bictegravir (BIC)
- Component 1: Arm 1.2: Doravirine (DOR) 100 mg q.d.: Women ≥ 20 weeks gestation not receiving TB drugs and receiving doravirine (DOR) 100 mg q.d., and their infants
  Interventions: Drug: Doravirine (DOR)
- Component 1: Arm 1.3: Tenofovir alafenamide (TAF) 10 mg q.d.: Women ≥ 20 weeks gestation not receiving TB drugs and receiving tenofovir alafenamide (TAF) 10 mg q.d. boosted with cobicistat, and their infants
  Interventions: Drug: Tenofovir alafenamide (TAF); Drug: Cobicistat
- Component 1: Arm 1.4: TAF 25 mg q.d. without boosting: Women ≥ 20 weeks gestation not receiving TB drugs and receiving TAF 25 mg q.d. without boosting, and their infants
  Interventions: Drug: Tenofovir alafenamide (TAF)
- Component 1: Arm 1.5: TAF 25 mg q.d. with boosting: Women ≥ 20 weeks gestation not receiving TB drugs and receiving TAF 25 mg q.d. boosted with cobicistat or ritonavir, and their infants
  Interventions: Drug: Tenofovir alafenamide (TAF); Drug: Cobicistat; Drug: Ritonavir
- Component 2: Arm 2.1: CAB LA: Women ≥ 24 weeks gestation who received at least one dose of long-acting injectable formulation of cabotegravir (CAB LA) any dose during pregnancy, and their infants
  Interventions: Drug: Cabotegravir (CAB)
- Component 3: Arm 3.1: Dolutegravir (DTG) 50 mg: Women ≥ 20 weeks gestation receiving first-line TB treatment with at least two of the following TB treatment drugs: isoniazid (INH), rifampin (RIF), rifabutin (RFB), ethambutol (EMB), pyrazinamide (PZA), moxifloxacin (MFX), and receiving dolutegravir (DTG) 50 mg twice daily (b.i.d.) when combined with RIF or 50 mg q.d. if RIF is not part of the TB regimen, and their infants
  Interventions: Drug: Dolutegravir (DTG); Drug: First-Line TB Treatment
- Component 3: Arm 3.2: ATV/r or DRV/r: Women ≥ 20 weeks gestation receiving first-line TB treatment with at least two of the following TB treatment drugs: isoniazid (INH), rifampin (RIF), rifabutin (RFB), ethambutol (EMB), pyrazinamide (PZA), moxifloxacin (MFX), and receiving atazanavir/ritonavir (ATV/r) ≥ 300/100 mg q.d. or darunavir/ritonavir (DRV/r) ≥ 600/100 mg b.i.d., and their infants
  Interventions: Drug: Atazanavir/ritonavir (ATV/r); Drug: Darunavir/ritonavir (DRV/r); Drug: First-Line TB Treatment
- Component 3: Arm 3.3: Lopinavir/ritonavir (LPV/r) 800/200 mg: Women ≥ 20 weeks gestation receiving first-line TB treatment with at least two of the following TB treatment drugs: isoniazid (INH), rifampin (RIF), rifabutin (RFB), ethambutol (EMB), pyrazinamide (PZA), moxifloxacin (MFX), and receiving lopinavir/ritonavir (LPV/r) 800/200 mg b.i.d., and their infants
  Interventions: Drug: Lopinavir/ritonavir (LPV/r); Drug: First-Line TB Treatment
- Component 4: Arm 4.1: Second-line TB treatment drugs: Women ≥ 20 weeks gestation receiving at least one of the following second-line TB treatment drugs, and their infants:
  * Levofloxacin (LFX) 750mg - 1000mg q.d.
  * Clofazimine (CFZ) 100mg q.d.
  * Linezolid (LZD) 300mg - 600mg q.d.
  * Bedaquiline (BDQ) 200mg three times per week (t.i.w.)
  * Delamanid (DLM) 100mg b.i.d.
  * Moxifloxacin (MFX) 400mg or 800mg q.d., and at least one other second-line TB treatment drug under study
  Interventions: Drug: Second-Line TB Treatment
- Component 5: Arm 5.1: ATV/r: Women post-delivery receiving ATV/r, and their infants
  Interventions: Drug: Atazanavir/ritonavir (ATV/r)
- Component 5: Arm 5.2: DRV/r: Women post-delivery receiving DRV/r, and their infants
  Interventions: Drug: Darunavir/ritonavir (DRV/r)
- Component 5: Arm 5.3: LPV/r: Women post-delivery receiving LPV/r, and their infants
  Interventions: Drug: Lopinavir/ritonavir (LPV/r)

INTERVENTIONS:
Drug: Bictegravir (BIC) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 1: Arm 1.1: Bictegravir (BIC) 50 mg q.d.
Drug: Tenofovir alafenamide (TAF) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 1: Arm 1.3: Tenofovir alafenamide (TAF) 10 mg q.d.; Component 1: Arm 1.4: TAF 25 mg q.d. without boosting; Component 1: Arm 1.5: TAF 25 mg q.d. with boosting
Drug: Cabotegravir (CAB) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 2: Arm 2.1: CAB LA
Drug: Dolutegravir (DTG) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 3: Arm 3.1: Dolutegravir (DTG) 50 mg
Drug: Atazanavir/ritonavir (ATV/r) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 3: Arm 3.2: ATV/r or DRV/r; Component 5: Arm 5.1: ATV/r
Drug: Darunavir/ritonavir (DRV/r) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 3: Arm 3.2: ATV/r or DRV/r; Component 5: Arm 5.2: DRV/r
Drug: Lopinavir/ritonavir (LPV/r) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 3: Arm 3.3: Lopinavir/ritonavir (LPV/r) 800/200 mg; Component 5: Arm 5.3: LPV/r
Drug: Cobicistat — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 1: Arm 1.3: Tenofovir alafenamide (TAF) 10 mg q.d.; Component 1: Arm 1.5: TAF 25 mg q.d. with boosting
Drug: Ritonavir — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 1: Arm 1.5: TAF 25 mg q.d. with boosting
Drug: First-Line TB Treatment — Participants will be receiving first-line TB treatment with at least two of the following TB treatment drugs: isoniazid (INH), rifampin (RIF), rifabutin (RFB), ethambutol (EMB), pyrazinamide (PZA), or moxifloxacin (MFX).
  Drugs will be administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants.
  Groups: Component 3: Arm 3.1: Dolutegravir (DTG) 50 mg; Component 3: Arm 3.2: ATV/r or DRV/r; Component 3: Arm 3.3: Lopinavir/ritonavir (LPV/r) 800/200 mg
Drug: Second-Line TB Treatment — Participants will be receiving second-line TB treatment with at least one of the following second-line TB treatment drugs:
  * Levofloxacin (LFX) 750mg - 1000mg q.d.
  * Clofazimine (CFZ) 100mg q.d.
  * Linezolid (LZD) 300mg - 600mg q.d.
  * Bedaquiline (BDQ) 200mg three times per week (t.i.w.)
  * Delamanid (DLM) 100mg b.i.d.
  * Moxifloxacin (MFX) 400mg or 800mg q.d., and at least one other second-line TB treatment drug under study
  Drugs will be administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants.
  Groups: Component 4: Arm 4.1: Second-line TB treatment drugs
Drug: Doravirine (DOR) — Administered consistent with the package inserts and/or instructions provided by the non-study sources who prescribe or supply the drugs to participants
  Groups: Component 1: Arm 1.2: Doravirine (DOR) 100 mg q.d.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) properties of antiretroviral (ARV) and anti-tuberculosis (TB) drugs administered during pregnancy and postpartum.

DETAILED DESCRIPTION:
This study will evaluate the pharmacokinetic (PK) properties of antiretroviral (ARV) and anti-tuberculosis (TB) drugs administered during pregnancy and postpartum.

IMPAACT 2026 is a Phase IV observational clinical study. Participants are not assigned to the drugs under study, but are already receiving the drugs for clinical care by prescription of their clinical care providers. They are enrolled into study arms according to the drugs they are receiving through clinical care, and if on multiple drugs of interest, are able to enroll into multiple arms simultaneously. No ARVs or TB treatment drugs are supplied as part of this study. All drugs under study are provided by non-study sources. The study sponsor added this observational study to an existing investigational new drug (IND) number for off-label use in case the participant's clinical care provider decides to prescribe a higher dose than the approved dose if the PK results for the approved dose indicate that drug exposure may be inadequate.

This study is comprised of five components which in turn are comprised of arms specific to each drug or drug combination being evaluated:

* Component 1 (Arms 1.1, 1.2. 1.3. 1.4. and 1.5): Pregnant women living with HIV (WLHIV) receiving oral ARVs and no TB drugs, and their infants.
* Component 2 (Arm 2.1): Pregnant WLHIV and HIV-uninfected women who received long-acting/extended release ARVs during pregnancy, and their infants.
* Component 3 (Arms 3.1, 3.2, and 3.3): Pregnant WLHIV receiving ARVs and first-line TB treatment, and their infants.
* Component 4 (Arm 4.1): Pregnant WLHIV and HIV-uninfected women receiving second-line TB treatment, and their infants.
* Component 5 (Arms 5.1, 5.2. and 5.3): Postpartum WLHIV breastfeeding while receiving oral ARVs, and their infants.

Each arm will open to accrual independently and will accrue independently over approximately 36 months from the first enrollment in each arm.

Participants in Component 1 will be followed up to 12 weeks after delivery for mothers and up to 24 weeks after birth for infants. Participants in Component 2 will be followed up to 5 weeks after delivery for mothers and infants. Participants in Components 3, 4, and 5 will be followed up to 24 weeks after delivery for mothers and infants.

Study visits may include:

* Component 1: Maternal clinical and laboratory evaluations and PK sampling at second trimester (2T), third trimester (3T), delivery, and 6-12 weeks post-partum (PP). Infant clinical evaluations and washout PK sampling at birth and 5-9 days after birth.
* Component 2: Maternal clinical and laboratory evaluations and PK sampling at delivery. Infant clinical evaluations and washout PK sampling at birth, 5-9 days, and 12-16 days after birth. Maternal and infant breast milk transfer PK sampling at 5-9 days, 12-16 days, and 3-5 weeks after delivery.
* Component 3: Maternal clinical and laboratory evaluations and PK sampling at second trimester (2T), third trimester (3T), delivery, and 2-8 weeks post-partum (PP). Infant clinical evaluations and washout PK sampling at birth and 5-9 days after birth. Maternal and infant breast milk transfer PK sampling at 5-9 days, 2-8 weeks, and 16-24 weeks after delivery.
* Component 4: Maternal clinical and laboratory evaluations and PK sampling at second trimester (2T), third trimester (3T), delivery, and 2-8 weeks post-partum (PP). Infant clinical evaluations and washout PK sampling at birth and 5-9 days after birth. Maternal and infant breast milk transfer PK sampling at 5-9 days, 2-8 weeks, and 16-24 weeks after delivery.
* Component 5: Maternal and infant clinical evaluations and breast milk transfer PK sampling at 5-9 days, 2-12 weeks, and 16-24 weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

Component 1: Pregnant WLHIV receiving oral ARVs and no TB drugs, and their infants

* Mother is of legal age or otherwise able to provide independent informed consent as determined by site standard operating procedures (SOPs) and consistent with site institutional review board (IRB)/ethics committee (EC) policies and procedures, and is willing and able to provide written informed consent for her own and her infant's participation in this study.
* Prior to study entry, HIV status confirmed as HIV infected per study protocol.
* At study entry, pregnant and in one of the following two enrollment windows based on best available obstetrical estimate of gestational age:

  * Second trimester: gestational age of 20 0/7 to 26 6/7 weeks
  * Third trimester: gestational age of 30 0/7 to 37 6/7 weeks
* At study entry, receiving at least one of the following oral ARV drugs or drug combinations, based on maternal report and available medical records:

  * Arm 1.1: Bictegravir (BIC) 50 mg q.d.
  * Arm 1.2: Doravirine (DOR) 100 mg q.d.
  * Arm 1.3: Tenofovir alafenamide (TAF) - 10 mg q.d. boosted with cobicistat
  * Arm 1.4: TAF 25 mg q.d. without boosting
  * Arm 1.5: TAF 25 mg q.d. boosted with cobicistat or ritonavir
* At study entry, planning to continue the current ARV regimen through at least 12 weeks post-delivery, based on maternal report and available medical records.
* At study entry, has been receiving the drug or drug combination under study at the required dose for at least two weeks, based on maternal report and available medical records.
* At study entry, assessed by study staff as having no identified barriers to completing initial PK sampling within 20 0/7 - 26 6/7 weeks gestation (second trimester) or 30 0/7 to 37 6/7 weeks gestation (third trimester) and within 14 days of enrollment.
* At study entry, if receiving a generic formulation of the drug or drug combination under study, approval of the formulation per study protocol.
* At study entry, not receiving any TB drugs (for either prophylaxis or treatment), based on maternal report and available medical records.

Component 2: Pregnant WLHIV and HIV-uninfected women who received long-acting/extended release ARVs during pregnancy, and their infants

* If of legal age or otherwise able to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures: Willing and able to provide written informed consent for her own and her infant's participation in this study.
* If not of legal age or otherwise unable to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures: Parent/guardian or other legally authorized representative of the mother and her infant is willing and able to provide written informed consent for the mother and her infant's study participation; in addition, when applicable, the mother is willing and able to provide written assent for her own and her infant's study participation.
* At study entry, intends to deliver at the study-affiliated clinic or hospital, based on maternal report.
* At study entry, gestational age of at least 24 0/7 weeks based on best available obstetrical estimate of gestational age, and not yet delivered.
* At study entry, has received at least one administration of the following, based on available medical records, during the current pregnancy:

  * Arm 2.1: Long-acting injectable formulation of cabotegravir (CAB LA) (any dose)

Component 3: Pregnant WLHIV receiving ARVs with first-line TB treatment, and their infants

* Mother is of legal age or otherwise able to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures, and is willing and able to provide written informed consent for her own and her infant's participation in this study.
* Prior to study entry, HIV status confirmed as HIV infected per study protocol.
* At study entry, pregnant and in one of the following two enrollment windows, based on best available obstetrical estimate of gestational age:

  * Second trimester: gestational age of 20 0/7 to 26 6/7 weeks
  * Third trimester: gestational age of 30 0/7 to 37 6/7 weeks
* At study entry, receiving at least two of the following first-line TB treatment drugs under study AND at least one of the following ARV drugs or drug combinations under study, based on maternal report and available medical records:

  * First-line TB treatment drugs:
  * Isoniazid (INH) 4-6 mg/kg (max 300 mg) q.d.
  * Rifampin (RIF) 8-12 mg/kg (max 600 mg) q.d.
  * Rifabutin (RFB) 150-300 mg q.d.
  * Ethambutol (EMB) 15-20 mg/kg q.d.
  * Pyrazinamide (PZA) 20-30 mg/kg q.d.
  * Moxifloxacin (MFX) 400 mg or 800mg q.d
  * ARVs:
  * Arm 3.1: Dolutegravir (DTG) 50 mg b.i.d. when combined with RIF or 50 mg q.d. if RIF is not part of the TB regimen
  * Arm 3.2: Atazanavir/ritonavir (ATV/r) ≥300/100 mg q.d. or Darunavir/ritonavir (DRV/r) ≥ 600/100 mg b.i.d.
  * Arm 3.3: Lopinavir/ritonavir (LPV/r) 800/200 mg b.i.d.
* At study entry, has been receiving the drug combination under study at the required dose for at least two weeks based on maternal report and available medical records.
* At study entry, assessed by study staff as having no identified barriers to completing initial PK sampling within 20 0/7 - 26 6/7 weeks gestation (second trimester) or 30 0/7 to 37 6/7 weeks gestation (third trimester) and within 14 days of enrollment.
* At study entry, if receiving a generic ARV or TB formulation of the drug or drug combination under study, approval of the formulation per study protocol.
* At study entry, planning to continue the current ARV regimen through at least 8 weeks post-delivery, based on maternal report and available medical records.

Component 4 Inclusion Criteria: Pregnant WLHIV and HIV-uninfected women receiving second-line TB treatment, and their infants

* Mother is of legal age or otherwise able to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures, and is willing and able to provide written informed consent for her own and her infant's participation in this study.
* Prior to study entry, HIV status confirmed as HIV-infected or HIV-uninfected, per study protocol.
* At study entry, pregnant and in one of the following two enrollment windows based on best available obstetrical estimate of gestational age:

  * Second trimester: gestational age of 20 0/7 to 26 6/7 weeks
  * Third trimester: gestational age of 30 0/7 to 37 6/7 weeks
* At study entry, receiving at least one of the following second-line TB treatment drugs under study, based on maternal report and available medical records:

  * Arm 4.1: Second-line TB treatment drugs:
  * Levofloxacin (LFX) 750mg - 1000mg q.d.
  * Clofazimine (CFZ) 100mg q.d.
  * Linezolid (LZD) 300mg - 600mg q.d.
  * Bedaquiline (BDQ) 200mg t.i.w.
  * Delamanid (DLM) 100mg b.i.d.
  * Moxifloxacin (MFX) 400mg or 800mg q.d and at least one other second-line TB treatment drug under study
* At study entry, has been receiving the drugs under study at the required dose for at least two weeks, based on maternal report and available medical records.
* At study entry, assessed by study staff as having no identified barriers to completing initial PK sampling within 20 0/7 - 26 6/7 weeks gestation (second trimester) or 30 0/7 to 37 6/7 weeks gestation (third trimester) and within 14 days of enrollment.
* At study entry, if receiving a generic formulation of the drug(s) under study, approval of the formulation per study protocol.

Component 5: Postpartum WLHIV breastfeeding while receiving oral ARVs, and their infants

* Mother is of legal age or otherwise able to provide independent informed consent as determined by site SOPs and consistent with site IRB/EC policies and procedures, and is willing and able to provide written informed consent for her own and her infant's participation in this study.
* Prior to study entry, HIV status confirmed as HIV infected, per study protocol.
* At study entry, within 5-9 days post-delivery (inclusive).
* At study entry, breastfeeding mother-infant pair intends to continue exclusive breastfeeding through at least 16 weeks post-delivery.
* At study entry, mother is receiving any of the following oral ARV drugs or drug combinations:

  * Arm 5.1: Atazanavir/ritonavir (ATV/r)
  * Arm 5.2: Darunavir/ritonavir (DRV/r)
  * Arm 5.3: Lopinavir/ritonavir (LPV/r)
* At study entry, mother has been receiving the drug(s) or drug combination(s) under study at the required dose for at least two weeks, based on maternal report and available medical records.
* At study entry, assessed by study staff as having no identified barriers to completing initial PK sampling within the 5-9 days post-delivery PK sampling window.
* At study entry, mother is planning to continue the current ARV regimen through at least 16 weeks post-delivery, based on maternal report and available medical records.
* At study entry, if receiving a generic ARV formulation of the drug or drug combination under study, approval of the formulation per study protocol.
* At study entry, infant weighs at least 1000 grams, based on available medical records.
* At study entry, infant does not have any severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the site investigator.

Components 1-4 Exclusion Criteria:

* At study entry, mother has received within the past 14 days medicines known to interfere with absorption, metabolism, or clearance of the drug or drug combination under study (see study protocol) based on maternal report and available medical records.

  * Note: RIF is permitted for mothers in Components 3 and 4 being evaluated for TB and ARV drug interactions.
* At study entry, has a clinical or laboratory finding or condition that, in the opinion of the site investigator, is likely to require a change of the ARV or TB drug under study during the period of study follow-up.
* Arms 1.3, 1.4 and 1.5 only: At study entry, mother has received TDF-based therapy within the past 6 months.

Component 5 Exclusion Criteria

* Mother is currently enrolled in Components 1, 2, 3, or 4.
* At study entry, the mother or infant has received within the past 14 days medicines known to interfere with absorption, metabolism, or clearance of the drug or drug combination under study based on maternal report and available medical records (see study protocol).
* At study entry, mother or infant has a clinical or laboratory finding or condition that, in the opinion of the site investigator, is likely to require a change of the drug under study during study follow-up.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant and postpartum women living with and without HIV (WLHIV and HIV-uninfected women) receiving ARV and/or TB drugs under study, and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Number of women who meet area under the curve (AUC) target in second trimester (2T) | Measured at 2T (20 0/7 weeks to 26 6/7 weeks of pregnancy)
  For Arms 1.1, and 1.2: BIC, DOR only
Number of women who meet area under the curve (AUC) target in third trimester (3T) | Measured at 3T (30 0/7 weeks to 37 6/7 weeks of pregnancy)
  For Arms 1.1, and 1.2: BIC, DOR only
Number of women who meet area under the curve (AUC) in postpartum (PP) | Measured at PP (6 to 12 weeks after delivery)
  For Arms 1.1, and 1.2: BIC, DOR only
Area under the curve (AUC) in second trimester (2T) | Measured at 2T (20 0/7 weeks to 26 6/7 weeks of pregnancy)
  For Arms 1.1, and 1.2: BIC, DOR only
Area under the curve (AUC) in third trimester (3T) | Measured at 3T (30 0/7 weeks to 37 6/7 weeks of pregnancy)
  For Arms 1.1, and 1.2: BIC, DOR only
Area under the curve (AUC) postpartum (PP) | Measured at PP (6 to 12 weeks after delivery)
  For Arms 1.1, and 1.2: BIC, DOR only
Tenofovir-diphosphate (TFV-DP) concentrations in peripheral blood mononuclear cells (PBMCs) and dried blood spots (DBS) in second trimester (2T) | Measured at 2T (20 0/7 weeks to 26 6/7 weeks of pregnancy)
  For Arms 1.3, 1.4, and 1.5 only
Tenofovir-diphosphate (TFV-DP) concentrations in peripheral blood mononuclear cells (PBMCs) and dried blood spots (DBS) in third trimester (3T) | Measured at 3T (30 0/7 weeks to 37 6/7 weeks of pregnancy)
  For Arms 1.3, 1.4, and 1.5 only
Tenofovir-diphosphate (TFV-DP) concentrations in peripheral blood mononuclear cells (PBMCs) and dried blood spots (DBS) postpartum (PP) | Measured at PP (6 to 12 weeks after delivery)
  For Arms 1.3, 1.4, and 1.5 only
Cord blood/maternal plasma concentration ratio at delivery | Measured on Day 0
  For Arm 2.1.: CAB only
Infant washout half-life after delivery (if not breastfeeding) | Measured on Day 0
  For Arm 2.1: CAB only
Maternal breast milk/maternal plasma concentration ratio (if breast feeding) | Measured at Day 0
  For Arm 2.1: CAB only
Infant plasma concentration at breast milk PK visit (if breast feeding) | Measured through Week 5
  For Arm 2.1: CAB only
Area under the curve (AUC) at second trimester (2T) | Measured at 2T (20 0/7 weeks to 26 6/7 weeks of pregnancy)
  For Arms 3.1, 3.2 and 3.3 only
Area under the curve (AUC) at third trimester (3T) | Measured at 3T (30 0/7 weeks to 37 6/7 weeks of pregnancy)
  For Arms 3.1, 3.2 and 3.3 only
Area under the curve (AUC) postpartum (PP) | Measured at PP (6 to 12 weeks after delivery)
  For Arms 3.1, 3.2 and 3.3 only
Area under the curve (AUC) at second trimester (2T) | Measured at 2T (20 0/7 weeks to 26 6/7 weeks of pregnancy)
  For Arm 4.1 only
Area under the curve (AUC) at third trimester (3T) | Measured at 3T (30 0/7 weeks to 37 6/7 weeks of pregnancy)
  For Arm 4.1 only
Area under the curve (AUC) postpartum (PP) | Measured at PP (6 to 12 weeks after delivery)
  For Arm 4.1 only
Maternal breast milk/maternal plasma concentration ratio | Measured through Week 24
  For Arms 5.1, 5.2, and 5.3 only
Infant plasma concentration | Measured through Week 24
  For Arms 5.1, 5.2, and 5.3 only

SECONDARY OUTCOMES:
Ratio of cord blood concentration to maternal blood concentration | Measured at Day 0
  For Components 1, 3 and 4, all Arms
Infant washout half-life of drug after birth (if the infant is not breastfeeding, and if the half-life is estimable) | Measured through Day 9
  For Components 1, 3 and 4, all Arms
Maternal breast milk/maternal plasma concentration ratio | Measured through Week 24
  For Components 3 and 4, if assessed
Infant plasma concentration | Measured through Week 24
  For Components 3 and 4, if assessed
Efavirenz, lopinavir, atazanavir, darunavir, dolutegravir, and/or raltegravir: AUC at second trimester (2T), third trimester (3T), and postpartum (PP) | Measured at Measured at 2T (20 0/7 to 26 6/7 weeks of pregnancy), 3T (30 0/7 to 37 6/7 weeks or pregnancy, and PP (2-8 weeks after delivery)
  For Component 4 only
Frequency of grade 3 or higher maternal adverse events | Measured through Week 24
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Frequency of grade 2 or higher infant adverse events | Measured through Week 24
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Frequency of maternal and infant serious adverse events | Measured through Week 24
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Frequency of grade 3 or higher maternal adverse events assessed as related to the drug under study | Measured through Week 24
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Frequency of grade 2 or higher infant adverse events assessed as related to the drug under study | Measured through Week 24
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Pregnancy outcome: occurrence of live birth versus fetal loss/stillbirth. | Measured on Day 0
Gestational age at birth | Measured on Day 0
Birth weight | Measured on Day 0
Occurrence of congenital anomaly | Measured from Day 0 through Week 24 for Components 1, 3, 4 and 5; measured from Day 0 through Week 5 for Component 2
Occurrence of mitochondrial disorder | Measured from Day 0 through Week 24 for Components 1, 3, 4 and 5; measured from Day 0 through Week 5 for Component 2
Number of infants with confirmed positive HIV nucleic acid test result | Measured from Day 0 through Week 24
  Determined according to diagnosis per local standard of care
Maternal HIV-1 RNA | Measured at 2T (20 0/7 to 26 6/7 weeks of pregnancy), 3T (30 0/7 to 37 6/7 weeks or pregnancy, and PP (2-12 weeks after delivery)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, MD, Study Chair — Boston University
Locations (23):
- United States (13):
  - Usc La Nichd Crs, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, San Diego, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - University of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV NICHD CRS, Miami, Florida
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Rush University Cook County Hospital Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS (Site ID: 4001), Chicago, Illinois
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
- Brazil (2):
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- Kenya Medical Research Institute / Walter Reed Project Clinical Research Center, Kericho CRS, Kericho, Kenya
- IMPAACT/ Gamma Project/ UPR Pediatric HIV/AIDS Research CRS, San Juan, Puerto Rico
- South Africa (3):
  - Wits RHI Shandukani Research, Johannesburg, Gauteng
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town
  - Famcru Crs, Tygerberg Hills
- Siriraj Hospital, Mahidol University NICHD CRS, Bangkok, Bangkoknoi, Thailand
- Baylor-Uganda CRS, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data

REFERENCES:
- [Derived] Powis KM, Pinilla M, McMorrow F, Stek A, Brooks KM, Shapiro DE, Knowles K, Eke AC, Greene E, Agwu A, Topete L, Browning R, Chakhtoura N, Arora P, Huang X, Best BM, Mirochnick M, Momper JD; IMPAACT 2026 Protocol Team. Pharmacokinetics and Safety of Bictegravir in Pregnant and Postpartum Persons With HIV and Their Infants. J Acquir Immune Defic Syndr. 2025 Mar 1;98(3):300-307. doi: 10.1097/QAI.0000000000003571. PMID 39813286